CLINICAL TRIAL: NCT01179997
Title: Tissue Doppler Imaging (TDI) Versus Electrocardiography (ECG) Interventricular Pacing Delay Optimization in Cardiac Resynchronization Therapy (CRT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacio Clinic Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, MD PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRT-opt
Record Dates: First submitted 2010-08-05; First posted 2010-08-11 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2010-05

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tissue Doppler Imaging (TDI) optimization (Active Comparator): Interventricular pacing delay optimized according to Tissue-Doppler echocardiography
  Interventions: Device: Interventricular pacing delay optimization by using Tissue Doppler-derived displacement curves
- Electrocardiographic optimization (Active Comparator): Interventricular pacing delay optimized according to QRS width observation in the 12-lead surface electrocardiogram
  Interventions: Device: Electrocardiographic optimization of the interventricular pacing delay according to QRS width

INTERVENTIONS:
Device: Interventricular pacing delay optimization by using Tissue Doppler-derived displacement curves
  Arms: Tissue Doppler Imaging (TDI) optimization
Device: Electrocardiographic optimization of the interventricular pacing delay according to QRS width
  Arms: Electrocardiographic optimization

SUMMARY:
The aim of this study was to compare the response to cardiac resynchronization therapy when the interventricular pacing interval was optimized by Tissue Doppler Imaging (TDI) to response when it was optimized following QRS width criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to de novo implant due to conventional cardiac resynchronization therapy indications.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)

PRIMARY OUTCOMES:
6-month echocardiographic response
  Reduction of the end-systolic volume (measured in mililiters according to transthoracic echocardiography) of >10% as compared to the baseline value.

SECONDARY OUTCOMES:
6-month clinical response
  Combined end-point consisting in no death due to cardiovascular reasons, no heart transplantation and distance increase of >10% (measured in meters) in the 6-minute walking test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Universitari, Barcelona, Catalonia, Spain